CLINICAL TRIAL: NCT00440206
Title: Multicenter Trial of Immunologic Markers to Predict Long Term Virologic Outcomes
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario HIV Treatment Network (Network)
Other Study IDs: 2002060-01H
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections
Keywords: HIV; Immune Markers
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Purpose is to identify whether immune markerscan predict success of salvage anti-retroviral therapy.

DETAILED DESCRIPTION:
Over the last several years two markers of disease have been utilized to determine if antiretroviral therapy has been successful, one is a CD4 cell count (reflects the immunocompetence of an infected individual) and a HIV viral load (a blood test used to determine the amount of HIV in the infected individual). However in patients who fail their first line of therapythe likelihood of extended resuppressing viral replication with subsequent therapies may be as low as 25-50%. This information may take several months to determine the new therapies possible continuing success. It would be preferable to have additional markers that respond to therapies in the first several weeks to such therapies, therfore possibly offering patients alternate treatment earlier without potentiatinglong term side effects and possible further drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV infected
* must be ≥18 years old
* must have been taking the same combination ARV regimen (≥3 drugs) for at least 3 months.
* Must be experiencing virologic failure (viral load ≥50 copies/mL on two occasions at least 2 weeks apart).
* must be changed to a salvage antiretroviral regimen
* Patient has to have signed and dated a full infomred consent.

Exclusion Criteria:

* Patient with any of the following abnormal laboratory test results in the previous 3 months:
* Hemaglobin <100 g/L
* Platelet count <20,000 cells/L
* INR ≥3.5 IU
* PTT ≥60 IU
* Patient with other significant underlying disease (non-HIV) that might impact immune markers ( eg. advanced liver disease, malignancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-09; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: J Angel, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - McMaster Health Science Center, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Maple Leaf Clinic, Toronto, Ontario
  - Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario